CLINICAL TRIAL: NCT05160727
Title: A Multicenter Phase II Clinical Study of Radiotherapy Combined With Tislelizumab and Irinotecan in MSS/pMMR Inoperable Recurrence and Metastatic Colorectal Cancer
Brief Title: Radiotherapy Combined With Tislelizumab and Irinotecan in MSS/pMMR Recurrence and Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ji Zhu, MD, Professor, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARTOnG-2104
Record Dates: First submitted 2021-11-16; First posted 2021-12-16 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Mismatch Repair-proficient; Colorectal Cancer Metastatic; Microsatellite Stable
Keywords: Tislelizumab; Irinotecan; colorectal cancer; mismatch repair-proficient; microsatellite stable
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tislelizumab; Irinotecan; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Concurrent Chemoradiotherapy:
  Radiation: The dose is determined according to the treatment site and the purpose of treatment.
  Irinotecan: 80mg/m2/w (UGT1A1*28 and *6: 6/6+GG) or 65mg/m2/w (UGT1A1*28 and *6: 6/7+GG or 6/6+GA) or 50mg/m2/w (UGT1A1*28 and *6: 7/7+GG or 6/6+AA or 6/7+GA) Tislelizumab: 200mg ivgtt d1 q3w
  Consolidation therapy: 2 weeks after the completion of chemoradiotherapy. Irinotecan: 200mg/m2 ivgtt d1 q3w. Tislelizumab: 200mg ivgtt d1 q3w. Efficacy assessment every 3 cycles.
  Interventions: Drug: Tislelizumab; Drug: Irinotecan; Radiation: radiotherapy

INTERVENTIONS:
Drug: Tislelizumab — 200mg ivgtt d1 q3w
Drug: Irinotecan — Concurrent Chemoradiotherapy:
  Irinotecan: 80mg/m2/w (UGT1A1*28 and *6: 6/6+GG) or 65mg/m2/w (UGT1A1*28 and *6: 6/7+GG or 6/6+GA) or 50mg/m2/w (UGT1A1*28 and *6: 7/7+GG or 6/6+AA or 6/7+GA) Consolidation therapy: 2 weeks after the completion of chemoradiotherapy. Irinotecan: 200mg/m2 ivgtt d1 q3w.
Radiation: radiotherapy — radiotherapy

SUMMARY:
Explore the efficacy of radiotherapy combined with Tislelizumab and irinotecan in MSS/pMMR inoperable recurrent and metastatic colorectal cancer patients; To evaluate the safety and tolerability of radiotherapy combined with Tislelizumab and irinotecan in MSS/pMMR inoperable recurrent and metastatic colorectal cancer; To evaluate the radiosensitization effects of Tslelizumab and irinotecan;

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of informed consent;
2. Aged 18-70 years old, regardless of gender;
3. Histologically confirmed as inoperable recurrent or metastatic colorectal adenocarcinoma;
4. Previously received oxaliplatin and fluorouracil based chemotherapy; No previous treatment with irinotecan;
5. NGS sequencing or immunohistochemistry prompts MSS/pMMR
6. At least one measurable lesion;
7. Palliative radiotherapy is required for clinical evaluation (except radiotherapy for bone or brain metastasis);
8. ECOG scores 0-2;
9. Expected survival ≥ 6 months;
10. The organ function of the patient was normal within 7 days before treatment, and the function of important organs met certain requirements.

Exclusion Criteria:

1. Pregnant or breastfeeding women;
2. There were primary lesions or metastases in the radiation field and had received radiotherapy before;
3. Previously received PD-1, PD-L1 or PD-L2 for any indication;
4. Those with other history of malignant disease in the past 5 years, except for cured skin cancer and cervical carcinoma in situ;
5. If there is an uncontrolled history of epilepsy, central nervous system disease or mental disorder, the investigator may determine that the clinical severity may hinder the signing of informed consent or affect the patient's oral medication compliance;
6. Clinically severe (ie, active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or more severe congestive heart failure or severe arrhythmia requiring medication intervention (see appendix 12), or a history of myocardial infarction in the last 12 months;
7. Organ transplantation requires immunosuppressive therapy Severe uncontrolled recurrent infections, or other serious uncontrolled concomitant diseases;
8. Subject blood routine and biochemical indicators do not meet the following criteria: hemoglobin ≥ 90g / L; absolute neutrophil count (ANC)≥ 1.5 × 109 / L; Alanine transaminase (ALT), aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal; alkaline phosphatase (ALP).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 18 weeks after treatment completion
  in radiation field

CONTACTS AND LOCATIONS:
Overall Officials: Ji Zhu, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No